CLINICAL TRIAL: NCT00390780
Title: A Comparative Randomized, Double-blind, Double-Dummy, Multicenter Study of the Efficacy and Safety of Miconazole Lauriad 50mg Administered Once a Day and Mycelex Troches (Clotrimazole 10mg) Administered Five Times a Day in the Treatment of Oropharyngeal Candidiasis in Immunocompromised Patients
Brief Title: Efficacy and Safety Study of Miconazole Lauriad to Treat Oropharyngeal Candidiasis in HIV Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BA/2004/01/04
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Results first posted 2013-08-29 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: Miconazole Lauriad; Oropharyngeal candidiasis; HIV patients; Mycology; Clinical picture of Oropharyngeal candidiasis; Candida culture positive; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Clotrimazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clotrimazole (Active Comparator): Clotrimazole troches, 10 mg, 5 times per day for 14 days
  Interventions: Drug: Clotrimazole
- miconazole Lauriad (Experimental): Miconazole Lauriad 50 mg mucoadhesive buccal tablet, once daily, for 14 days
  Interventions: Drug: miconazole Lauriad

INTERVENTIONS:
Drug: miconazole Lauriad — 50 mg buccal tablet once a day for 14 days
  Arms: miconazole Lauriad
Drug: Clotrimazole — 10mg troches administered Five Times a Day for 14 days
  Arms: Clotrimazole

SUMMARY:
The purpose of this study is to evaluate the clinical cure of miconazole Lauriad 50 mg (1x50mg) Bioadhesive buccal tablets compared with clotrimazole troches (5x10mg) after 14 days of treatment (at the test of cure visit, at Day 17-19).

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical picture of oropharyngeal candidiasis
* Confirmation of oropharyngeal candidiasis by candida culture positive
* HIV-positive patients
* Patients 18 years of age

Exclusion Criteria:

* Patients with signs or symptoms of systemic candidiasis
* Patients with signs or symptoms of esophagitis
* Pregnant or breast-feeding women
* Patients who have taken systemic antifungals within the past 30 days
* Patients who have taken local antifungals within the past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (21):
  - University of Alabama, Department of diagnostic Sciences School of Dentistry, Birmingham, Alabama
  - L.A. Gay & Lesbian center, Health & Mental, health services, Los Angeles, California
  - East Bay AIDS Center, Oakland, California
  - 1401 Noth Palm Canyon, Palm Springs, California
  - University of Connecticut, School of dental medicine, Farmington, Connecticut
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Fort Lauderdale, Florida
  - Ryan White Title III Clinic, LaBelle, Florida
  - University of Miami, Miami, Florida
  - Triple O Medical Services, West Palm Beach, Florida
  - Department of oral medicine and diagnostic sciences UIC college of dentistry, Chicago, Illinois
  - Plus Clinic, University of Maryland Dental school, Baltimore, Maryland
  - Henry Ford Hospital and Wayne State University, Division of infectious diseases, Detroit, Michigan
  - AIDS Community Research Initiative of America, New York, New York
  - Department Diagnostics Sciences, UNC, Chapel Hill, North Carolina
  - East Carolina University, Brody School of Medicine, Greenville, North Carolina
  - University of Oklahoma, College of medicine, Tulsa, Oklahoma
  - Lehigh Valley Hospital Clinical Research Department of Medicine, Allentown, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Bering Omega Dental Clinic, Houston, Texas
  - Eastern Virginia Medical Center, Center for comprehensive care of immune deficiency, Norfolk, Virginia
- Canada (6):
  - Downtown Infectious Disease Clinic, Vancouver, British Columbia
  - Providence Health Center British Columbia Centre for excellence in HIV/AIDS, Vancouver, British Columbia
  - Health Sciences Center, Winnipeg, Manitoba
  - University of Ottawa Health Services, Ottawa, Ontario
  - Montreal Chest Institutes immunodeficiency clinic, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 25 July 06 to 27 December 07 A total of 30 clinical sites (private practice and hospitals) in US, Canada and South Africa screened patients for this study, and 28 sites randomized patients
Pre-assignment Details: There were no significant events or approaches following participant enrollment and prior to group assignment
Groups:
- Miconazole Lauriad Buccal Tablet: Miconazole Lauriad 50 mg mucoadhesive buccal tablet, once daily, for 14 days
- Clotrimazole Troches: Clotrimazole troches, 10 mg, 5 times per day, for 14 days
Period: Overall Study
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Started | 291 | 287
Treatment | 290 (One patient randomized to miconazole lost study drug, never started treatment, and was discontinued.) | 287
Completed | 268 | 260
Not Completed | 23 | 27
Not completed — Not completed | 10 | 4
Not completed — Protocol Violation | 6 | 4
Not completed — Lost to Follow-up | 3 | 6
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Inclusion criteria not satisfied | 0 | 2
Not completed — Lost to follow up and other reasons | 0 | 1
Not completed — Investigator decision, SAE, other reason | 0 | 1
Not completed — SAE, death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Clotrimazole Troches: Clotrimazole troches, 10 mg, 5 times per day for 14 days
- Total: Total of all reporting groups
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches | Total
Number analyzed (Participants) | 290 | 287 | 577
Age Continuous [Mean (Full Range); unit: years] | 37.5 (9.7) [18 to 73] | 36.5 (9.1) [18 to 72] | 37.0 (9.4) [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 168 | 341
  Male | 117 | 119 | 236
Region of Enrollment [Number; unit: participants]
  United States | 67 | 62 | 129
  Canada | 3 | 3 | 6
  South Africa | 220 | 222 | 442

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure (Defined as a Complete Resolution of Signs and Symptoms) After 14 Days of Treatment at the Test of Cure Visit (Day 17-Day 22) Using Murray Scoring Scale
Description: Murray scoring scale range: extent of oral lesions (signs) 0 (none) to 3 (extensive or confluent), ordinal; symptoms (soreness/burning) 0 (absent) to 3 (severe), ordinal. Clinical cure was defined as a complete resolution of signs and symptoms (extent of oral lesions score = 0, symptoms score = 0). Clinical failure was defined as any patient who failed to be clinically cured by the treatment.
Time Frame: 17 to 22 days
Population: Intent-to-Treat (ITT, all randomized patients who took at least 1 dose of study medication)
  Per Protocol (PP, all patients in ITT without major protocol deviation, with positive fungal culture, completed at least 10 days of treatment, had main efficacy criteria at test of cure, compliant within 71.4% to 120%, and no forbidden medications taken)
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants
  Clinical Cure-ITT | 176 | 187
  Clinical Failure-ITT | 114 | 100
  Clinical Cure-PP | 164 | 175
  Clinical Failure-PP | 76 | 61
Statistical Analysis 1: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Analyses for ITT and PP populations: H0: clinical cure rate for miconazole Lauriad minus clinical cure rate for clotrimazole troches is less than or equal to -0.15 H1: clinical cure rate for miconazole Lauriad minus clinical cure rate for Mycelex troches is greater than -0.15; Test type: Non-Inferiority or Equivalence — Non inferiority assumptions: Type of test: one-sided Inferiority margin: -15% Expected cure rate: 70% Type I error: 2.5% Type II error: 5%; p > 0.025, one-sided test — Significance level was <0.025; comparison of proportion clinical cure = 0.15, 95% CI 1-sided [lower limit -0.15]

2. Secondary Outcome: Clinical Cure at Day 7 (Using Murray Scoring Scale)
Description: as for outcome 1
Time Frame: 7 days
Population: ITT (all randomized patients who took at least 1 dose of study medication)
  PP (all patients in ITT without major protocol deviation, with positive fungal culture, completed at least 10 days of treatment, had main efficacy criteria at test of cure, compliant within 71.4% to 120%, and no forbidden medications taken)
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants
  Clinical Cure-ITT | 67 | 71
  Clinical Failure-ITT | 210 | 202
  Data Missing-ITT | 13 | 14
  Clinical Cure-PP | 60 | 63
  Clinical Failure-PP | 180 | 173
Statistical Analysis 1: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Analysis for ITT and PP populations: H0: clinical cure rate for miconazole Lauriad minus clinical cure rate for clotrimazole troches is less than or equal to -0.15 H1: clinical cure rate for miconazole Lauriad minus clinical cure rate for Mycelex troches is greater than -0.15; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > 0.025, one-sided noninferiority test — Significance level was <0.025; comparison of proportion clinical cure = 0.15, 95% CI 1-sided [lower limit -0.15]

3. Secondary Outcome: Clinical Success at Test-of-cure Visit (Day 17-22) (Using Murray Scoring Scale)
Description: Murray scoring scale range: extent of oral lesions (signs) 0 (none) to 3 (extensive or confluent), ordinal; symptoms (soreness/burning) 0 (absent) to 3 (severe), ordinal. Clinical success was defined as clinical cure or clinical improvement. Clinical cure was defined as a complete resolution of signs and symptoms (extent of oral lesions score = 0, symptoms score = 0). Clinical improvement was defined as having no visible lesion (extent of lesions score = 0) and minimal symptoms (soreness/burning score <2). Clinical failure was defined as any patient who failed to be clinically cured by the treatment.
Time Frame: 17 to 22 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants
  Clinical Success-ITT | 188 | 199
  Clinical Failure-ITT | 80 | 61
  Data Missing-ITT | 22 | 27
  Clinical Failure-PP | 67 | 51
  Clinical Success-PP | 173 | 185
Statistical Analysis 1: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Analysis for ITT population: H0: clinical success rate for miconazole Lauriad minus clinical success rate for clotrimazole troches is less than or equal to -0.15 H1: clinical success rate for miconazole Lauriad minus clinical success rate for Mycelex troches is greater than -0.15; Test type: Non-Inferiority or Equivalence — Non inferiority assumptions: Type of test: one-sided Inferiority margin: -15% Type I error: 2.5% Type II error: 5%; p = 0.0974, Cochran-Mantel-Haenszel — Significance level was <0.025; compare proportion of clinical success = 0.15, 95% CI 1-sided [lower limit -0.15]
Statistical Analysis 2: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Analysis for PP population: H0: clinical success rate for miconazole Lauriad minus clinical success rate for clotrimazole troches is less than or equal to -0.15 H1: clinical success rate for miconazole Lauriad minus clinical success rate for Mycelex troches is greater than -0.15; Test type: Non-Inferiority or Equivalence — Non inferiority assumptions: Type of test: one-sided Inferiority margin: -15% Type I error: 2.5% Type II error: 5%; p = 0.1115, Cochran-Mantel-Haenszel — Significance level was <0.025; Compare proportion of clinical success = 0.15, 95% CI 1-sided [lower limit -0.15]

4. Secondary Outcome: Clinical Success at Day 7 (Using Murray Scoring Scale)
Description: as for outcome 3
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants
  Clinical Success-ITT | 92 | 89
  Clinical Failure-ITT | 185 | 184
  Data Missing-ITT | 13 | 14
  Clinical Success-PP | 82 | 78
  Clinical Failure-PP | 158 | 158
Statistical Analysis 1: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — Non inferiority assumptions: Type of test: one-sided Inferiority margin: -15% Type I error: 2.5% Type II error: 5%; p = 0.8787, Cochran-Mantel-Haenszel — Significance level was <0.025; compare proportion of clinical success = 0.15, 95% CI 1-sided [lower limit -0.15]
Statistical Analysis 2: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; [analysis description as in outcome 3, analysis 2]; Test type: Non-Inferiority or Equivalence — Non inferiority assumptions: Type of test: one-sided Inferiority margin: -15% Type I error: 2.5% Type II error: 5%; p = 0.7969, Cochran-Mantel-Haenszel — Significance level was <0.025; compare proportion of clinical success = 0.15, 95% CI 1-sided [lower limit -0.15]

5. Secondary Outcome: Partial Response at Test of Cure Visit (Days 17-22) Using Murray Scoring Scale
Description: Murray scoring scale range: extent of oral lesions (signs) 0 (none) to 3 (extensive or confluent), ordinal; symptoms (soreness/burning) 0 (absent) to 3 (severe), ordinal. Clinical success was defined as clinical cure or clinical improvement. Partial response is having decrease in Murray extent of oral lesions score by at least 1 level and a stable Murray symptoms score, with partial symptom response defined as having a decrease in the Murray symptoms (soreness/burning) score by at least 1 level and a stable Murray extent of oral lesions score, and partial clinical/symptom response defined as decrease in Murray extent of oral lesions score by at least 1 level and a decrease in the Murray symptoms (soreness/burning) score by at least 1 level
Time Frame: 17 to 22 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants
  Partial response-ITT | 139 | 140
  Partial response-PP | 120 | 123
Statistical Analysis 1: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Analysis for ITT population: H0: partial response rate for miconazole Lauriad minus partial response rate for clotrimazole troches is less than or equal to -0.15 H1: partial response rate for miconazole Lauriad minus partial response rate for Mycelex troches is greater than -0.15; Test type: Non-Inferiority or Equivalence — Non inferiority assumptions: Type of test: one-sided Inferiority margin: -15% Type I error: 2.5% Type II error: 5%; p = 0.8820, Cochran-Mantel-Haenszel — Significance level was <0.025; compare proportion of partial response = 0.15, 95% CI 1-sided [lower limit -0.15]
Statistical Analysis 2: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Analysis for PP population: H0: partial response rate for miconazole Lauriad minus partial response rate for clotrimazole troches is less than or equal to -0.15 H1: partial response rate for miconazole Lauriad minus partial response rate for Mycelex troches is greater than -0.15; Test type: Non-Inferiority or Equivalence — Non inferiority assumptions: Type of test: one-sided Inferiority margin: -15% Type I error: 2.5% Type II error: 5%; p = 0.9033, Cochran-Mantel-Haenszel — Significance level was <0.025; compare proportion of partial response = 0.15, 95% CI 1-sided [lower limit -0.15]

6. Secondary Outcome: Mycological Cure at the Test of Cure Visit (Day 17-22)
Description: Mycological cure was defined as a patient who had "no yeast isolated" when oral specimens were cultured for fungi.
Time Frame: 17 to 22 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants
  Mycological Cure-ITT | 79 | 71
  Mycological Failure-ITT | 185 | 185
  Data Missing-ITT | 26 | 31
  Mycological Cure-PP | 73 | 64
  Mycological Failure-PP | 164 | 168
Statistical Analysis 1: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Test type: Non-Inferiority or Equivalence — Non-inferiority statistical analysis for ITT population; p = 0.5816, Chi-squared — Significance level was <0.025; difference in proportion mycologic cure = 0.15, 95% CI 1-sided [lower limit -0.15]
Statistical Analysis 2: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Test type: Non-Inferiority or Equivalence — Non-inferiority statistical analysis for PP population; p = 0.4439, Chi-squared — Significance level was <0.025; difference in proportion mycologic cure = 0.15, 95% CI 1-sided [lower limit -0.15]

7. Secondary Outcome: Relapse at the Late Post-Therapy Visit (Day 35-38)
Description: "Number of patients" represents the number of participants who completed visit 6 (the late post-therapy visit on Days 35-38) and had been a clinical success at test-of-cure visit (visit 5). For this subset of participants, relapse was defined as a patient who responded to treatment by clinical cure or improvement (i.e., "clinical success") on Days 17-22 at the test-of-cure visit (visit 5) and subsequently had an increase in the extent of oral lesions or symptoms, as assessed at the late post-therapy visit on Days 35-38 (visit 6). No relapse indicates participants who were considered a "clinical success" at visit 5 and did not have a subsequent increase in the extent of oral lesions or symptoms, as assessed at the late post-therapy visit (visit 6). The remaining number of participants in the Intent-to-Treat population who did not meet the criteria for relapse assessment at visit 6 is listed under "Not Analyzed-ITT".
Time Frame: 35 to 38 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants
  Number of patients-ITT | 183 | 197
  Relapse-ITT | 51 | 53
  No relapse-ITT | 132 | 144
  Not Analyzed-ITT | 107 | 90
  Number of patients-PP | 168 | 184
  Relapse-PP | 45 | 49
  No relapse-PP | 123 | 135
Statistical Analysis 1: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Test type: Non-Inferiority or Equivalence — Non-inferiority statistical analysis for ITT population; p = 0.8330, Chi-squared — Significance level is <0.025; difference in proportion relapsed = 0.15, 95% CI 1-sided [lower limit -0.15]
Statistical Analysis 2: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Test type: Non-Inferiority or Equivalence — Non-inferiority statistical analysis for PP population; p = 0.9738, Chi-squared — Significance level is <0.025; difference in proportion relapsed = 0.15, 95% CI 1-sided [lower limit -0.15]

8. Secondary Outcome: Oral Discomfort Using Visual Analog Scale (VAS)
Description: Visual analog scale was used by the patient in the patient diary. The scale ranged from 0 (no oral discomfort) to 10 (maximum oral discomfort)
Time Frame: 14 days
Population: Intent-to-Treat (ITT, all randomized patients who took at least 1 dose of study medication)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
units on a scale | 0.8 [0 to 9] | 0.4 [0 to 6]

9. Secondary Outcome: General and Local Tolerability and Oral Discomfort
Description: Overall local adverse reactions, including gingival inflammation, gum pain, alterations in taste of food when eating, alterations in taste when not eating, and dry mouth. Visit 4 occurred on Day 14.
Time Frame: 14 days
Population: Safety Population (same as ITT population, includes all randomized patients who took at least one dose of the study medication)
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants
  Gingival Inflammation-Visit 4 (R canine fossa) | 34 | 26
  No Gingival Inflammation-Visit 4 (R canine fossa) | 235 | 233
  Data Missing (Inflammation)-Visit 4 (R fossa) | 21 | 28
  Gingival Inflammation-Visit 4 (L canine fossa) | 30 | 24
  No Gingival Inflammation-Visit 4 (L canine fossa) | 239 | 236
  Data Missing (Inflammation)-Visit 4 (L fossa) | 21 | 27
  Gum Pain-Visit 4 | 32 | 24
  No Gum Pain-Visit 4 | 240 | 236
  Data Missing (Gum Pain)-Visit 4 | 18 | 27
  Taste of Food Alteration-Visit 4 | 63 | 54
  No Taste of Food Alteration-Visit 4 | 209 | 206
  Data Missing (Taste of Food Alteration)-Visit 4 | 18 | 27
  Taste When Not Eating Alteration-Visit 4 | 63 | 52
  No Taste When Not Eating Alteration-Visit 4 | 209 | 208
  Data Missing (Taste When Not Eating)-Visit 4 | 18 | 27
  Dry Mouth-Visit 4 | 57 | 67
  No Dry Mouth-Visit 4 | 215 | 193
  Data Missing (Dry Mouth)-Visit 4 | 18 | 27

10. Secondary Outcome: Duration of Adhesion of Miconazole Lauriad 50 mg Mucoadhesive Buccal Tablet
Description: The mean durations of adhesion from initiation of treatment to Day 14 of miconazole Lauriad 50 mg mucoadhesive buccal tablet (or, in the case of the Clotrimazole troches treatment arm, the placebo mucoadhesive buccal tablet) were rounded to the nearest hour
Time Frame: 14 days
Population: ITT (all randomized patients who took at least 1 dose of study medication)
Measure: Mean (Full Range); unit: hours
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
hours | 13 [0 to 14] | 13 [0 to 14]

11. Secondary Outcome: Systemic Exposure of Miconazole Lauriad 50 mg Bioadhesive Buccal Tablet
Description: Number of patients with detectable plasma concentration at Visit 3 (day 7)
Time Frame: 7 days
Population: ITT (all randomized patients who took at least 1 dose of study medication)
Measure: Number; unit: participants
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants | 0 | 0

12. Secondary Outcome: Susceptibility of Candida Species by Microdilution Test
Description: minimum inhibitory concentration (MIC) in nonresponders at test-of-cure visit
Time Frame: Initiation of treatment to Day 17 to 22
Population: ITT (all randomized patients who took at least 1 dose of study medication), nonresponders (participants with progression to a higher visible lesion extent score or no reduction in oral lesion extent score at the test of cure [Day 17 to 22] visit)
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
mcg/ml
  Clotrimazole MIC for C. albicans (n=9, 7) | 0.0099 (0.0040) | 0.0073 (0.0039)
  Miconazole MIC for C. albicans (n=9, 7) | 0.0764 (0.0995) | 0.1664 (0.3679)
Statistical Analysis 1: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Analysis for Clotrimazole minimum inhibitory concentration (MIC) between treatment groups; Test type: Superiority or Other; p = 0.1860, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Miconazole Lauriad Buccal Tablet vs Clotrimazole Troches; Analysis for Miconazole minimum inhibitory concentration (MIC) between treatment groups; Test type: Superiority or Other; p = 0.9564, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Treatment Compliance
Description: Number of patients who were 100% compliant with the treatment regimen
Time Frame: Initiation of treatment to Day 14
Population: ITT (all randomized patients who took at least 1 dose of study medication)
Measure: Number; unit: participants compliant
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Number analyzed (Participants) | 290 | 287
participants compliant | 253 | 250

ADVERSE EVENTS:
Time Frame: 14 days study treatment, then 21 days of follow-up
Arm/Group | Miconazole Lauriad Buccal Tablet | Clotrimazole Troches
Serious Adverse Events (participants affected / at risk) | 10/290 | 9/287
Other Adverse Events (participants affected / at risk) | 85/290 | 84/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Miconazole Lauriad Buccal Tablet (N=290) | Clotrimazole Troches (N=287)
AIDS dementia complex (Infections and infestations) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Retroviral infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Shigella infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Miconazole Lauriad Buccal Tablet (N=290) | Clotrimazole Troches (N=287)
Diarrhea (Gastrointestinal disorders) | 26 (30) | 23 (28)
Nausea (Gastrointestinal disorders) | 19 (25) | 22 (28)
Vomiting (Gastrointestinal disorders) | 11 (11) | 9 (10)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 5 (5)
Gastroenteritis (Infections and infestations) | 4 (4) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 7 (7)
Headache (Nervous system disorders) | 22 (25) | 19 (23)
Ageusia (Nervous system disorders) | 7 (9) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 5 (6)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Fatigue (General disorders) | 8 (9) | 6 (7)
Pain (General disorders) | 3 (3) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
GGT increased (Investigations) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less